CLINICAL TRIAL: NCT06058130
Title: Combination of Antiplatelet and Anticoagulation for Acute Ischemic Stroke Patients Witn Concomitant Non-valvular Atrial Fibrillation and Extracranial/Intracranial Artery Stenosis
Brief Title: Combination of Antiplatelet and Anticoagulation for AIS Patients Witn Concomitant NVAF and Extracranial/Intracranial Artery Stenosis
Acronym: ALLY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ALLY
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-09

CONDITIONS: Acute Ischemic Stroke; Atrial Fibrillation; Stenosis, Carotid; Intracranial Atherosclerosis
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Carotid Stenosis; Intracranial Arteriosclerosis | interventions — Anticoagulants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticoagulation alone (Active Comparator): Rivaroxaban 20mg once daily or 15mg once daily / Dabigatran 110mg twice daily or 150mg twice daily
  Interventions: Drug: Anticoagulant Oral
- Anticoagulation combined with antiplatelet therapy (Experimental): Rivaroxaban 20mg once daily or 15mg once daily or 10mg once daily / dabigatran 110mg twice daily or 150mg twice daily+ aspirin 100mg once daily / clopidogrel 75mg once daily / ticagrelor 90mg twice daily / cilostazol 100mg twice daily
  Interventions: Drug: Anticoagulation combined with antiplatelet therapy

INTERVENTIONS:
Drug: Anticoagulant Oral — Anticoagulation alone
  Arms: Anticoagulation alone
Drug: Anticoagulation combined with antiplatelet therapy — Anticoagulation combined with antiplatelet therapy
  Arms: Anticoagulation combined with antiplatelet therapy

SUMMARY:
The goal of this clinical trial is to compare the safety and effectiveness of anticoagulation combined with antiplatelet therapy in acute ischemic stroke (AIS) patients with concomitant non-valvular atrial fibrillation (NVAF) and extracranial/intracranial artery stenosis. Participants will be 1:1 randomized into anticoagulation alone or anticoagulation combined with antiplatelet therapy. The primary endpoint is composite events 3 months after enrollment.

DETAILED DESCRIPTION:
Concomitant NVAF and extracranial/intracranial artery stenosis will greatly increase the risk of stroke, even with standard anticoagulation. However, clinicians may be concerned with the high risk of bleeding complications of anticoagulation combined with antiplatelet therapy. The goal of this clinical trial is to evaluate the safety and effectiveness of anticoagulation combined with antiplatelet therapy in acute ischemic stroke (AIS) patients with concomitant non-valvular atrial fibrillation (NVAF) and extracranial/intracranial artery stenosis. Participants will be 1:1 randomized into anticoagulation alone or anticoagulation combined with antiplatelet therapy. The primary endpoint is composite events 3 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Acute ischemic stroke or TIA with onset < 7 days
* Have a history or newly diagnosed as NVAF
* Concomitant stenosis (>50%) of carotid artery/intracranial artery, of which the ischemic lesion located within the territory

Exclusion Criteria:

* Chronic renal dysfunction (GFR < 30ml/min) or severe hepatic injury
* Have a history or newly diagnosed as valvular heart disease
* Mural thrombus in heart
* Contraindications of anticoagulation or antiplatelet therapy, e.g. severe intracranial hemorrhage
* Myocardial infarction within 6 months before enrollment or received percutaneous coronary intervention in the past
* Have or plan to receive CEA or CAS in the following 3 months
* Life expectancy less than 1 year
* Plan to receive invasive surgery in the following 3 months and have high risk of uncontrollable bleeding
* Pregnant or lactating women
* Individuals identified by researchers as unsuitable for participation in the study due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2171 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The rate of 90-day Composite events | 90 days
  Composite events including ischemic stroke, hemorrhagic stroke, myocardial infarction, systemic embolism, major extracranial hemorrhage, and vascular death within 90 days after enrollment

SECONDARY OUTCOMES:
The rate of 90-day ischemic stroke | 90 days
  Ischemic stroke within 90 days after enrollment
The rate of 90-day hemorrhagic stroke | 90 days
  Hemorrhagic stroke within 90 days after enrollment
The rate of 90-day myocardial infarction | 90 days
  Myocardial infarction within 90 days after enrollment
The rate of 90-day systemic embolism | 90 days
  Systemic embolism within 90 days after enrollment
The rate of 90-day major extracranial hemorrhage | 90 days
  Major extracranial hemorrhage within 90 days after enrollment
The rate of 90-day non-major bleeding | 90 days
  Non-major bleeding within 90 days after enrollment
The rate of 90-day vascular death | 90 days
  Vascular death within 90 days after enrollment
The rate of 90-day all-cause death | 90 days
  All-cause death within 90 days after enrollment
Discharge modified Rankin scale score | At discharge, an average of 7 days
  Modified Rankin scale (mRS) at discharge. MRS ranges from 0 to 6, with a higher score indicating worse functional outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Jiaxing Second Hospital, Jiaxing

IPD SHARING:
Plan to Share IPD: No